CLINICAL TRIAL: NCT04787289
Title: A Comparison of 2 Standard Doses of Bevacizumab in Combination With Chemotherapy in Epithelial Ovarian Cancer - a Pragmatic Trial
Brief Title: A Comparison of 2 Standard Doses of Bevacizumab in Combination With Chemotherapy in Epithelial Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Jenny Ko, Medical Oncologist, British Columbia Cancer Agency
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEV-DOSE
Record Dates: First submitted 2021-03-01; First posted 2021-03-08 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Cancer; Platinum-resistant Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Higher Standard dosing as per standard regimen (Active Comparator): bevacizumab 15mg/kg + chemotherapy
  Interventions: Drug: Bevacizumab
- Lower standard dosing bevacizumab plus chemotherapy (Experimental): bevacizumab 7.5mg/kg + chemotherapy
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Low standard dose of bevacizumab, combined with single agent chemotherapy (7.5mg/kg IV Q3w or 5mg/kg IV Q2w)

SUMMARY:
A pragmatic, two armed, study comparing 2 standard doses of an anti-cancer drug called bevacizumab, given in combination with Chemotherapy. The study will be offered to ovarian cancer patients whose disease is platinum chemotherapy resistant . Higher doses of anti-cancer based drugs are not always better than lower doses and can cause more side effects without improvement of cancer. These patients will be randomly assigned either 7.5 mg/kg or 15mg/kg of bevacizumab combined with chemotherapy . Comparing these two doses will determine if the lower dose-level is non-inferior, and could lead to practice changes.

DETAILED DESCRIPTION:
Study team proposes to compare 2 standard doses of an anti-cancer drug called bevacizumab, 7.5mg/kg per dose vs. 15mg/kg per dose, given in combination with chemotherapy in patients with ovarian cancer that progressed on platinum chemotherapy. Higher doses in cases of antibody-based drugs like bevacizumab are not always better than lower doses, and in fact can cause more side effects without improving survival or shrinkage of cancer. Both 7.5 and 15mg/kg doses of bevacizumab every 3 weeks are used as standard protocol in BC Cancer for ovarian cancer patients, but only 15mg/kg doses are allowed for patients with ovarian cancer that progressed on platinum chemotherapy. This study is a pragmatic two-arm blinded study in which 70 patients with platinum-resistant ovarian cancer and eligible for bevacizumab + chemotherapy will be randomly assigned either to lower or higher standard dose of bevacizumab , combined with chemotherapy. Treating clinicians will decide how long the treatment will continue per standard of care. Duration of cancer control on CT scans, side effect profiles, and quality of life related to the two arms will be compared. If demonstrated, this finding will be practice-changing, with comparable efficacy and quality of life, potentially improved safety profile, as well as reduced provincial drug costs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of epithelial ovarian cancer, primary peritoneal, or fallopian tube carcinoma according to WHO Classification of tumours that is advanced/metastatic/recurrent or unresectable and for which no curative therapy exists.
* Platinum resistant disease (progression within six months of completing a platinum-containing protocol). In this case, progression from the last line of therapy would be defined as radiologic progression by RECIST 1.1 criteria on CT or MR.
* Presence of clinically and/or radiologically documented disease. All radiology studies must be performed within 28 days of randomization.
* All patients must have measurable disease as defined by RECIST 1.1. The criteria for defining measurable disease are as follows:

  * Chest x-ray > 20 mm
  * CT scan (with slice thickness of 5 mm) > 10 mm longest diameter
  * Physical exam (using calipers) > 10 mm Lymph nodes by CT scan > 15 mm measured in short axis
* Patients must be >= 18 years of age.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Any number of prior lines of treatment is permitted. However, all patients must have received at least one prior regimen of chemotherapy including platinum. All patients may have received other therapies including immunotherapy, hormone therapy, or PARP inhibitors.
* Patients must have never received an anti-angiogenesis inhibitor including bevacizumab.
* A BC Cancer "Compassionate Access Program" (CAP) request must be approved prior to treatment
* Radiation: prior external beam radiation is permitted provided a minimum of 28 days (4 weeks) have elapsed between the last dose of radiation and date of treatment initiation. Exceptions may be made for low-dose, non-myelosuppressive radiotherapy after consultation with sponsor.
* Surgery: Previous surgery is permitted provided that a minimum of 28 days (4 weeks) have elapsed between any major surgery and date of randomization/registration, and that wound healing has occurred.
* Women of childbearing potential must have agreed to use a highly effective contraceptive method during the study and for up to 5 months after the last dose of chemotherapy/bevacizumab. A woman is considered to be of "childbearing potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgical sterility defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation, or vasectomy/vasectomized partner.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to any study specific procedures (see Section 6.0) to document their willingness to participate.

Patients who cannot give informed consent (i.e. mentally incompetent patients, or those physically incapacitated such as comatose patients) are not to be recruited into the study. Patients competent but physically unable to sign the consent form may have the document signed by their Legally Acceptable Representative (LAR) or legal guardian. Each patient will be provided with a full explanation of the study before consent is requested.

* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits. Investigators must assure themselves the patients registered on this trial will be available for complete documentation of the treatment, response assessment, adverse events, and follow-up.

Exclusion Criteria:

* Patients with a history of other active or current malignancies that require active treatment.
* Patients with serious illness or medical conditions that might be aggravated by treatment or limit compliance including, but not limited to:

  * History of significant neurologic or psychiatric disorder which would impair the ability to obtain consent or limit compliance with study requirements.
  * Uncontrolled hypertension
  * Active uncontrolled or serious infection (viral, bacterial or fungal)
  * Other medical conditions that might be aggravated by study treatment
* Patients receiving concurrent treatment with other anti-cancer therapy or investigational agents.
* Neutrophils less than 1 x 10^9 /L
* Pregnancy or breastfeeding
* Bleeding diathesis
* History of bowel obstruction or unresolved bowel obstruction (refer to the BC Cancer protocols above)
* Uncontrolled arterial or venous thromboembolism (note: once controlled, patient may still be eligible).
* Myocardial infarction (MI) or cerebrovascular accident (CVA) within 4 months.
* Untreated or uncontrolled central nervous system (CNS) metastatic disease.
* Open, non-healing wounds or known fistulas that have not healed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 years months
  duration of time from registration to time progression

SECONDARY OUTCOMES:
Overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 years months
  duration of time from registration to time of death from any cause.
Duration of response | From time of objective response until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 years months
  Duration of response
Compare treatment-emergent grade 3-5 AEs | 4 months after last dose
  Compare treatment-emergent grade 3-5 AEs
Quality of Life changes | during treatment and 4 weeks after coming off treatment
  Quality of Life changes
Estimate drug cost savings | through study completion, up to 4 years
  Estimate drug cost savings

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Ko, Principal Investigator — BC Cancer
Locations (2):
- Canada (2):
  - Abbotsford Centre, BC Cancer Agency, Abbotsford, British Columbia
  - BC Cancer - Vancouver, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No